CLINICAL TRIAL: NCT04684992
Title: Telehealth Administration of 13C-Spirulina Gastric Emptying Breath Test (13C-GEBT) Usability Study
Brief Title: GEBT Telehealth Administration Usability Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairn Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PRO-CD-046
Record Dates: First submitted 2020-12-08; First posted 2020-12-28 (Actual); Results first posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-07

CONDITIONS: Gastroparesis
Keywords: Gastroenterology; Gastric emptying breath test; Telehealth
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- GEBT Telehealth Administration Usability (Experimental): Establish the usability of a telehealth platform for the administration of GEBT
  Interventions: Device: GEBT Telehealth Administration Usability

INTERVENTIONS:
Device: GEBT Telehealth Administration Usability — Establish the usability of a telehealth platform for the administration of GEBT

SUMMARY:
The purpose of this study is to establish the usability of a telehealth platform for the administration of GEBT.

DETAILED DESCRIPTION:
This study is intended to demonstrate that the 13C-Spirulina Gastric Emptying Breath Test (GEBT) can be successfully administered via a telehealth platform. Telehealth administration of GEBT is where a trained Cairn employee uses a video link to remotely supervise the completion of the test request form, collection of breath samples, cooking and consumption of the test meal and return of breath samples by the patient to Cairn.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, greater than or equal to 18 years of age at the time of signing the consent form, from healthy and intended use population (i.e. symptomatic for gastroparesis). Women of childbearing potential must not be pregnant at the time of GEBT administration.
* Ability to eat test meal and provide breath samples
* Access to a microwave oven at home
* Internet connection and telehealth accessible device (smart phone/tablet/computer with visual and voice capability) at home
* Environment to sit comfortably and quietly at home

Exclusion Criteria:

* History or physical exam suggestive of systemic disease such as pathophysiologic disorders such as renal failure, chronic heart disease, chronic respiratory disease, liver disease, or malabsorption syndrome
* History of abdominal surgery except appendectomy
* Females on hormone replacement therapy other than birth control medications
* Receipt of any investigational drug within 4 weeks of the study
* Pregnancy
* Intolerance or allergy to any component of GEBT meal
* History of neurological or psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex Ryder, MD, PhD, Principal Investigator — Cairn Diagnostics
Locations (1):
- Cairn Diagnostics, Brentwood, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | GEBT Telehealth Administration Usability
Started | 36
Completed | 34
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | GEBT Telehealth Administration Usability
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Patient Ability to Prepare and Administer the 13C-Spirulina GEBT, Under the Supervision of a Telehealth Professional, According to Instructions
Description: Ability to prepare GEBT will be assessed by the telehealth administrator's observation of the patient.
Time Frame: 1 day
Measure: Number; unit: participants
Arm/Group | GEBT Telehealth Administration Usability
Number analyzed (Participants) | 34
participants
  Transfer meal to cooking cup without spilling | 34
  Remove oxygen absorber | 34
  Added correct amount of water | 34
  Egg meal cooked for correct length of time | 34
  Egg flipped middle of cooking | 34
  Egg appeared adequately cooked | 34

2. Primary Outcome: Patient Ability to Prepare and Administer the 13C-Spirulina GEBT, Under the Supervision of a Telehealth Professional, According to Instructions
Description: Ability to prepare GEBT will be assessed by a patient questionnaire.
Time Frame: up to 1 week
Population: Study participants assessed on a patient questionnaire whether the meal preparation instructions were clear and easy to follow.
Measure: Number; unit: participants
Arm/Group | GEBT Telehealth Administration Usability
Number analyzed (Participants) | 34
participants | 34

3. Primary Outcome: Patient Ability to Complete the GEBT Test Request Form, Under the Supervision of a Telehealth Professional, According to the Instructions
Description: Ability to complete the GEBT test request form will be assessed by Cairn accessioning personnel upon receipt of returned breath samples.
Time Frame: 2-4 days
Measure: Number; unit: participants
Arm/Group | GEBT Telehealth Administration Usability
Number analyzed (Participants) | 34
participants
  Test Request Form returned with samples | 34
  Patient Information Entered Correctly | 33
  Pre-meal sample times recorded | 33
  Meal start/end times recorded correctly | 34
  Post-meal sample times recorded | 34

4. Primary Outcome: Patient Ability to Complete the GEBT Test Request Form, Under the Supervision of a Telehealth Professional, According to the Instructions
Description: Ability to complete the GEBT test request form will be assessed by a patient questionnaire.
Time Frame: up to 1 week
Population: Participants assessed easy of completing the GEBT test request form.
Measure: Number; unit: participants
Arm/Group | GEBT Telehealth Administration Usability
Number analyzed (Participants) | 34
participants | 34

5. Primary Outcome: Patient Ability to Collect GEBT Breath Samples Under the Supervision of a Telehealth Professional
Description: Ability to collect GEBT breath samples will be assessed by examination of GEBT results for participants (ensuring adequate CO2 in each sample/delta values follow expected pattern if collected in correct order).
Time Frame: up to 1 week
Measure: Number; unit: participants
Arm/Group | GEBT Telehealth Administration Usability
Number analyzed (Participants) | 34
participants
  Telehealth administrator observed condensate | 33
  Post meal samples collected within 5 minutes | 33
  Clinical lab personnel observed condensate | 34
  Adequate %CO2 (>1%) | 34
  Samples follow excretion curve shape | 34
  Breath samples easy to collect | 34

6. Primary Outcome: Ability to Successfully Ship Kits/Breath Samples to/From Home
Description: Ability to ship GEBT kits/breath samples to/from home will be assessed by surveying patients regarding shipping and by recording the dates that kits were shipped and received
Time Frame: Up to 3 weeks
Measure: Number; unit: participants
Arm/Group | GEBT Telehealth Administration Usability
Number analyzed (Participants) | 34
participants
  Kit arrived before test administration | 34
  Breath samples received within 28-days | 34

7. Primary Outcome: Ability of a Telehealth Platform to Function Correctly
Description: Verification that the software is user friendly and not subject to frequent failures during use will be assessed by a telehealth administrator questionnaire
Time Frame: 1 day
Measure: Number; unit: participants
Arm/Group | GEBT Telehealth Administration Usability
Number analyzed (Participants) | 34
participants
  No platform issues? | 32
  No lost connection? | 32
  No text reminder issues? | 31

8. Primary Outcome: Ability of a Telehealth Platform to Function Correctly
Description: Verification that the software is user friendly and not subject to frequent failures during use will be assessed by a patient questionnaire
Time Frame: Up to 3 weeks
Population: Participants assessed reliability and ease of use of telehealth platform.
Measure: Number; unit: participants
Arm/Group | GEBT Telehealth Administration Usability
Number analyzed (Participants) | 34
participants | 32

9. Primary Outcome: Safety of Telehealth Administration of 13C-Spirulina GEBT Versus Administration in a Clinician's Facility
Description: Any adverse events reported will be reviewed by Cairn's medical director to assess that there is no more than expected frequency of adverse events during administration of GEBT by a telehealth professional than would be expected during administration of GEBT in a clinician's facility. This will be performed by comparing the current rate of events in a physician's office versus under the supervision of a telehealth professional as identified through the risk analyses performed for GEBT administration.
Time Frame: Up to 3 weeks
Population: There were no adverse events associated with telehealth administration via the telehealth procedure (e.g., burns during microwave cooking or injuries from breath collection apparatus).
Measure: Number; unit: AEs associated with telehealth
Arm/Group | GEBT Telehealth Administration Usability
Number analyzed (Participants) | 34
AEs associated with telehealth | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | GEBT Telehealth Administration Usability
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 3/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GEBT Telehealth Administration Usability (N=34)
Excessive burping and nausea (Gastrointestinal disorders) | 1
Severe bloating and excessive gas (Gastrointestinal disorders) | 1
Vomiting and dehydration (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/92/NCT04684992/Prot_000.pdf